CLINICAL TRIAL: NCT06164275
Title: A Phase II Multi-Center Open-Label Trial of Six Doses of Pembrolizumab Monotherapy Prior to Limited Chemotherapy as Front-Line Therapy for Patients With Classical Hodgkin Lymphoma, Including Elderly Patients.
Brief Title: Pembrolizumab Followed by Chemotherapy for the Treatment of Patients With Classical Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 23H06; NCI-2023-08756 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00219738; NU 23H06 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2023-11-29; First posted 2023-12-11 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Classic Hodgkin Lymphoma
MeSH Terms: interventions — Biopsy; Specimen Handling; Dacarbazine; Doxorubicin; pembrolizumab; Magnetic Resonance Spectroscopy; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Pembrolizumab and AVD) (Experimental): INDUCTION: Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Treatment repeats repeat every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo disease assessment. Patients with a response complete 3 additional cycles of pembrolizumab, undergo disease assessment and proceed to consolidation. Patients without response or with progressive disease proceed to consolidation.
  CONSOLIDATION: Patients receive doxorubicin IV, vinblastine IV and dacarbazine IV on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity for 2 to 6 cycles dependent upon response and disease type. Patients undergo echocardiography/MUGA scan, CT scan, PET scan and blood sample collection throughout the study and may undergo tumor biopsy during screening.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Dacarbazine; Drug: Doxorubicin; Procedure: Echocardiography; Procedure: Multigated Acquisition Scan; Biological: Pembrolizumab; Procedure: Positron Emission Tomography; Drug: Vinblastine

INTERVENTIONS:
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Dacarbazine — Given IV
  Other Names: 4-(Dimethyltriazeno)imidazole-5-carboxamide; 5-(Dimethyltriazeno)imidazole-4-carboxamide; Asercit; Biocarbazine; Dacarbazina; Dacarbazina Almirall; Dacarbazine - DTIC; Dacatic; Dakarbazin; Deticene; Detimedac; DIC; Dimethyl (triazeno) imidazolecarboxamide; Dimethyl Triazeno Imidazol Carboxamide; Dimethyl Triazeno Imidazole Carboxamide; dimethyl-triazeno-imidazole carboxamide; Dimethyl-triazeno-imidazole-carboximide; DTIC; DTIC-Dome; Fauldetic; Imidazole Carboxamide; Imidazole Carboxamide Dimethyltriazeno; WR-139007
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; MUGA; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; Keytruda; Lambrolizumab; MK-3475; Pembrolizumab Biosimilar BCD-201; SCH 900475
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Drug: Vinblastine — Given IV
  Other Names: Vincaleucoblastine; VLB

SUMMARY:
This phase II trial tests how well giving pembrolizumab followed by chemotherapy with doxorubicin, vinblastine and dacarbazine works to treat patients with classical Hodgkin lymphoma. Pembrolizumab is a type of drug called a "monoclonal antibody (mAb)" that uses the body's immune system to help fight and kill cancer cells. Chemotherapy drugs, such as doxorubicin, vinblastine and dacarbazine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing or by stopping them from spreading. Giving pembrolizumab followed by chemotherapy may work to treat patients with classical Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the percent of patients that achieve a complete response (CR) after frontline pembrolizumab monotherapy induction, among classic Hodgkin lymphoma (cHL) patients with early unfavorable or advanced stage disease, per Lugano 2014 response criteria at positron emission tomography (PET) #2.

SECONDARY OBJECTIVES:

I. To assess the efficacy of a reduced number of cycles (2-4) of doxorubicin (adriamycin), vinblastine, and dacarbazine (AVD) when used following treatment with frontline pembrolizumab monotherapy in classic Hodgkin lymphoma (cHL), per Lugano 2014 Response Criteria.

II. To assess the safety and tolerability of sequential immunotherapy with upfront pembrolizumab followed by AVD chemotherapy in cHL per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (ver.) 5.0.

III. To assess progression-free-survival (PFS) of cHL patients who received sequential immunotherapy with upfront pembrolizumab followed by AVD chemotherapy, assessed by central review, according to Lugano 2014 Response Criteria.

IV. To assess overall survival (OS) of cHL patients who received sequential immunotherapy with upfront pembrolizumab followed by AVD chemotherapy.

V. To assess the CR rate at the end of pembrolizumab (PEM) induction by PET-computed tomography (CT) in all treated patients, regardless of number of cycles of PEM received, per Lugano 2014 Response Criteria.

OUTLINE:

INDUCTION: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 of each cycle. Treatment repeats repeat every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo disease assessment. Patients with a response complete 3 additional cycles of pembrolizumab, undergo disease assessment and proceed to consolidation. Patients without response or with progressive disease proceed to consolidation.

CONSOLIDATION: Patients receive doxorubicin IV, vinblastine IV and dacarbazine IV on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity for 2 to 6 cycles dependent upon response and disease type. Patients undergo echocardiography/ multigated acquisition (MUGA) scan, CT scan, PET scan and blood sample collection throughout the study and may undergo tumor biopsy during screening.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 1 year, and every 6 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of Ann Arbor Stage III or IV classic Hodgkin lymphoma (cHL) or Ann Arbor Stage I and Stage II classic Hodgkin lymphoma with at least one unfavorable risk factor by National Comprehensive Cancer Network (NCCN) criteria.

NCCN Unfavorable Factors include bulky disease defined as:

* A mass >10 cm disease in any dimension or
* Mediastinal mass ratio greater than one third defined as maximum width of mediastinal ass/intrathoracic diameter at T5-6
* B symptoms
* Erythrocyte sedimentation rate (ESR) ≥ 50
* And >3 sites of disease

  * Patients must have measurable fludeoxyglucose (FDG)-avid disease by Lugano 2014 response criteria
  * Patients must have previously untreated disease
  * Patients must be age ≥ 18 years
  * Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 per evaluation performed within 7 days prior to the date of the first dose of study intervention
  * Leukocytes (WBC) ≥ 3,000/mcL unless attributed to neoplastic involvement of the bone marrow
* Platelet transfusions are acceptable prior to treatment to achieve the above numbers, however growth factors are not allowed within 14 days of registration
* No lower limit if cytopenia is related to bone marrow involvement.

  * Absolute neutrophil count (ANC) ≥ 500/mcL unless attributed to neoplastic involvement of the bone marrow
* Platelet transfusions are acceptable prior to treatment to achieve the above numbers, however growth factors are not allowed within 14 days of registration
* No lower limit if cytopenia is related to bone marrow involvement

  * Hemoglobin (Hgb) ≥ 8 g/dL unless attributed to neoplastic involvement of the bone marrow
* Platelet transfusions are acceptable prior to treatment to achieve the above numbers, however growth factors are not allowed within 14 days of registration
* No lower limit if cytopenia is related to bone marrow involvement

  * Platelets (PLT) ≥ 25,000/mcL unless attributed to neoplastic involvement of the bone marrow
* Platelet transfusions are acceptable prior to treatment to achieve the above numbers, however growth factors are not allowed within 14 days of registration
* No lower limit if cytopenia is related to bone marrow involvement

  * Total bilirubin ≤1.5 × institutional upper limit of normal (ULN) OR direct bilirubin ≤ institutional ULN for participants with total bilirubin levels >1.5 × institutional ULN
  * Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) ≤ 2.5 x institutional ULN

    ≤ 5 × institutional ULN for participants with liver metastases
  * Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x institutional ULN

    ≤ 5 × institutional ULN for participants with liver metastases
  * Creatinine OR measured or calculated creatinine clearance (CrCl) (Glomerular filtration rate [GFR] can also be used in place of creatinine or CrCl) ≤ 1.5 x institutional ULN or ≥ 30 mL/min for participant including for participants with creatinine levels > 1.5 × institutional ULN
* Creatinine clearance (CrCl) should be calculated per institutional standard

  * International normalized ratio (INR) or prothrombin (PT) or partial thromboplastin time (aPTT) ≤ 1.5 × institutional ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
  * Patients of child-bearing potential (POCBP) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from time of informed consent, for the duration of study participation, and for 120 days following completion of therapy. POCBP must not donate eggs as per timelines for use of contraception. Should a POCBP become pregnant or suspect they are pregnant while they or their partner is participating in this study, POCBP should inform their treating physician immediately.

NOTE: A POCBP is any person with an egg-producing reproductive tract (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy
* Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)

  * Patients with sperm-producing reproductive capacity (PWSPRC) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from time of informed consent, for the duration of study participation, and for 120 days following completion of therapy. PWSPRC treated or enrolled on this protocol must also agree to refrain from donating sperm, from time of informed consent, for the duration of study participation, and for 120 days following completion of therapy
  * POCBP must have a negative pregnancy test within 7 days prior to registration on study NOTE: a negative urine pregnancy test is also required within 72 hours (3 days) prior to first dose of pembrolizumab and therefore may need to be repeated if screening test is more than 72 hours (3 days) prior to the first dose. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
  * Patients must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Diagnosis of nodular lymphocyte-predominant Hodgkin lymphoma
* Patients who have had prior systemic chemotherapy, radiation therapy, immunotherapy, or other systemic therapy (including investigational agents) for the treatment of cHL.

NOTE: If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy. No radiation therapy for Hodgkin lymphoma (cHL) will be allowed prior to and while participation on this clinical trial, including for system control

* Patients who are actively participating in a clinical trial with an investigational agent or device or has participated in a clinical trial with an investigational agent or device within 30 days of the anticipated treatment start date.

NOTE: Patients who have entered the follow-up phase of an investigational study will be eligible to participate as long as ≥ 30 days has elapsed since the administration of the last dose of an investigational treatment for a disease/condition other than cHL

* Patients who have known active central nervous system (CNS) metastases and/or lymphomatous meningitis are not eligible
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab, and/or any of its excipients
* Patients who have any contraindication to the use of any of the chemotherapeutic agents used in this study
* Patients who have had an allogenic tissue or solid organ transplant
* Patients who are pregnant or nursing NOTE: Pregnant persons are excluded from this study because the chemotherapy regimen (AVD) includes adriamycin (also known as doxorubicin), which is an anthracycline; anthracyclines are known chemotherapy agents with the potential for teratogenic or abortifacient effects. In addition, the investigational agent, pembrolizumab, has the potential for embryo-fetal toxicity. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with adriamycin (doxorubicin) as part of the AVD chemotherapy regimen, and the investigational agent, pembrolizumab, breastfeeding should be discontinued if the mother is treated with AVD and/or pembrolizumab.
* Patients who have a diagnosis of immunodeficiency or are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to registration are not eligible. NOTE: Replacement therapy (e.g., thyroxine, insulin, physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed
* Patients who have a known history of active TB (Bacillus Tuberculosis) are not eligible
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Symptomatic congestive heart failure (ejection fraction lower than institutional lower limit of normal [LLN]
  * Unstable angina pectoris
  * Cardiac arrhythmia
* Patients who have any prior malignancy OR a known additional malignancy that is progressing or requires active treatment are not eligible. NOTE: Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer. Participants with low-risk early-stage prostate cancer (T1-T2a, Gleason score ≤ 6, and PSA < 10 ng/mL) either treated with definitive intent or untreated in active surveillance with stable disease are not excluded
* Patients who have active autoimmune disease that has required systemic treatment in the past 2 years are not eligible (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs) NOTE: Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed
* Patients who have a history of (non-infectious) pneumonitis that required steroids or current pneumonitis are not eligible
* Patients who have an active infection requiring systemic therapy are not eligible, except for uncomplicated urinary tract infections
* Patients are not eligible who have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Patients who have known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial are not eligible
* Patients may not be pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, from registration through 120 days after the last dose of trial treatment
* Patients who have received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4, anti-OX-40 or anti-LAG-3 agent are not eligible
* Patients who have a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) are not eligible NOTE: HIV testing is not required unless mandated by local health authority
* Patients who have an active hepatitis B (e.g., hepatitis B surface antigen [HbsAg] reactive) or hepatitis C (e.g. hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected) are not eligible. NOTE: Testing for hepatitis B or C is not required unless mandated by local health authority
* Patients requiring urgent tumor debulking
* Patients who received a live vaccine within 30 days of planned start of study therapy are not eligible. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, some varicella/zoster vaccines, yellow fever, rabies, bacillus calmette-guerin (BCG), and typhoid vaccine.

NOTE: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed. Coronavirus 19 (COVID-19) vaccines for injection are generally messenger RNA vaccines and are also allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of complete response (CR) | Up to 5 years
  Assessed by position emission tomography (PET)-computed tomography (CT). CR defined as 1-3 on the five-point scale per Lugano (Lugano 2014 Response Criteria). Patients with 1-3 per Deauville criteria will be considered a complete response. Response will be determined, using a proportion and an exact binomial 95% confidence interval.

SECONDARY OUTCOMES:
Efficacy of reduced cycles of treatment with doxorubicin (adriamycin) vinblastine, doxorubicin (AVD) for patients with CR | Up to 5 years
  Patients that are identified as CR will be treated with AVD for 2-4 cycles and are evaluated again. Similarly, CR rate will be determined using a proportion and an exact binomial 95% confidence interval.
Incidence of adverse events | Up to 5 years
  Frequency and severity of adverse events by type, severity (grade), timing, and attribution to pembrolizumab will be assessed according to the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Overall survival (OS) | From start of treatment administration per protocol until death, up to 5 years
  Kaplan Meier curves will be used and 6-month, 1-year, and 2-year OS if applicable, will be calculated.
Progression free survival (PFS) | From the start of treatment administration per protocol until the first occurrence of disease relapse, progression, re-initiation of cytotoxic chemotherapy, or death due to disease, up to 5 years
  Kaplan Meier curves will be used and 6-month, 1-year, and 2-year PFS if applicable, will be calculated.
Assess the CR rate at the end of PEM induction by PET-CT i | Up to 5 years
  The CR rate at the end of the PEM treatment, using a proportion and an exact binomial 95% confidence interval, will be estimated for all patients that were treated with PEM.

CONTACTS AND LOCATIONS:
Overall Officials: Jane N Winter, MD, Principal Investigator — Northwestern University
Locations (4):
- United States (4):
  - Stanford Cancer Center, Stanford, California
  - Northwestern University, Chicago, Illinois
  - Northwestern Delnor IL258, Geneva, Illinois
  - Cadence Health - CDH, Warrenville, Illinois